CLINICAL TRIAL: NCT01497613
Title: Personalized Reminder Information and Social Management System - PRISM
Brief Title: A Personalized Reminder Information and Social Management System
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sara J Czaja, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20100482
Record Dates: First submitted 2011-12-13; First posted 2011-12-22 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Social Isolation; Social Support (Formal and Informal); Well-being/Quality of Life
Keywords: Socialization; Well-being; Quality of Life; Connectivity
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRISM B: Notebook Condition (Active Comparator): Telephone check-in calls and a notebook containing similar categories of information as the features on the PRISM C computer system such as a resource guide; games; classroom and information, calendar.
  Interventions: Behavioral: PRISM B: Notebook Condition
- PRISM C: Computer Condition (Experimental): A computer-based system designed to support socialization and access to resources; knowledge and prospective memory. The system is placed in the homes of those randomized to the condition for 12 months.
  Interventions: Behavioral: PRISM C: Computer Condition

INTERVENTIONS:
Behavioral: PRISM C: Computer Condition — A specialized computer system designed to support social connectivity and access to resources; knowledge and prospective memory
  Arms: PRISM C: Computer Condition
Behavioral: PRISM B: Notebook Condition — Telephone check-in calls and a notebook that contains information about community resources, games; topics of interests to seniors; a calendar and contact list.
  Arms: PRISM B: Notebook Condition

SUMMARY:
Although technology offers great potential for enhancing the health and well-being of older adults, robust studies are needed to quantify the value of technology and further the investigators understanding of barriers to technology access among older adults and of strategies that are effective in removing these barriers. This cross-site randomized field trial will evaluate a simple to use Personalized Reminder Information and Social Management System (PRISM) designed to support social connectivity, memory, skill building and resource access for older adults. The PRISM system (PRISM C condition) will be compared to an notebook information control condition (PRISM B condition). The target population is older adults who live at home alone and are at risk for isolation. The goal of the study is to gather systematic evidence about the value of technology for older adults and to identify factors that affect use and usability, acceptance and technology adoption. The investigators will also gather longitudinal data on the benefits of the system. Participants aged 65 - 85 years (100 per site) will be randomly assigned following baseline assessment to one of two conditions: PRISM C condition where participants receive the technology system or the PRISM B condition only control where participants receive a notebook that includes information similar to that provided in PRISM C (e.g., resource guide). The categories of information provided in the notebook is similar to the features provided on the system. Participants will include males and females who do not have a home computer and who have limited Internet experience. The intervention period is 12 months. A battery of measures that includes demographic information, attitudes towards technology (including computer self-efficacy and computer comfort), technology, computer and Internet experience, functional independence and well-being, emotional well-being social support/isolation, and quality of life will be administered at baseline, and 6 and 12 months post randomization. In addition, the investigators will assess cognitive abilities at baseline and twelve months. The investigators will also gather data regarding technology use and social interactions via a brief telephone interview at 18 months post randomization.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years
* Live alone in the community in an independent residence
* Minimum computer and Internet use in the past three months
* English speaking
* Able to read English at the 6th grade level
* Has a telephone
* 20/60 Vision with or without correction
* Not employed or volunteering more than 5 hrs/week
* Does not spend more than 10 hrs./week at a Senior Center or Formal organization
* Planning to remain in the area in same living arrangements for duration of intervention period

Exclusion Criteria:

* Blind or deaf
* Cognitively impaired (MMSE) < 26
* Fuld Object Memory Test < 20 or 19
* Terminal illness
* Severe motor impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J. Czaja, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Boot WR, Charness N, Czaja SJ, Sharit J, Rogers WA, Fisk AD, Mitzner T, Lee CC, Nair S. Computer proficiency questionnaire: assessing low and high computer proficient seniors. Gerontologist. 2015 Jun;55(3):404-11. doi: 10.1093/geront/gnt117. Epub 2013 Oct 9. PMID 24107443
- [Background] Czaja SJ, Boot WR, Charness N, A Rogers W, Sharit J, Fisk AD, Lee CC, Nair SN. The personalized reminder information and social management system (PRISM) trial: rationale, methods and baseline characteristics. Contemp Clin Trials. 2015 Jan;40:35-46. doi: 10.1016/j.cct.2014.11.004. Epub 2014 Nov 8. PMID 25460342
- [Background] Yoon JS, Charness N, Boot WR, Czaja SJ, Rogers WA. Depressive Symptoms as a Predictor of Memory Complaints in the PRISM Sample. J Gerontol B Psychol Sci Soc Sci. 2019 Jan 10;74(2):254-263. doi: 10.1093/geronb/gbx070. PMID 28575476
- [Background] Mitzner TL, Rogers WA, Fisk AD, Boot WR, Charness N, Czaja SJ, Sharit J. Predicting Older Adults' Perceptions about a Computer System Designed for Seniors. Univers Access Inf Soc. 2016 Jun;15(2):271-280. doi: 10.1007/s10209-014-0383-y. Epub 2014 Sep 7. PMID 31186624
- [Result] Czaja SJ, Boot WR, Charness N, Rogers WA, Sharit J. Improving Social Support for Older Adults Through Technology: Findings From the PRISM Randomized Controlled Trial. Gerontologist. 2018 May 8;58(3):467-477. doi: 10.1093/geront/gnw249. PMID 28201730
- [Derived] Mitzner TL, Savla J, Boot WR, Sharit J, Charness N, Czaja SJ, Rogers WA. Technology Adoption by Older Adults: Findings From the PRISM Trial. Gerontologist. 2019 Jan 9;59(1):34-44. doi: 10.1093/geront/gny113. PMID 30265294

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Started | 150 | 150
Completed | 113 | 131
Not Completed | 37 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.34 (7.4) | 76.97 (7.3) | 76.15 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 119 | 234
  Male | 35 | 31 | 66
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change in Social Isolation Measured by Friendship Scale
Description: Measures the level of social isolation from baseline to 6th month follow-up. Lower score means less social isolation. Range (0-24) .
Time Frame: Baseline and 6th month
Population: Some participants did not complete the questionnaire. 149 participants from PRISM B and 133 from PRISM C contributed to at least one of the two time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 149 | 133
units on a scale
  Baseline | 18.75 (4.1) | 19.72 (3.7)
  6th month follow-up: number analyzed (Participants) | 118 | 133
  6th month follow-up | 18.94 (4.3) | 20.27 (3.7)

2. Primary Outcome: Change in Level of Social Support Measured by Social Support Scale
Description: Measures the level of social support from baseline to 6th month follow-up. Higher score means more social support. Range (6-36).
Time Frame: Baseline and 6th month
Population: Some participants did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 150 | 150
units on a scale
  Baseline | 24.90 (6.9) | 25.33 (6.9)
  6th month follow-up: number analyzed (Participants) | 119 | 134
  6th month follow-up | 23.98 (6.9) | 26.12 (7.2)

3. Primary Outcome: Change Overall Well-being Measured by SF-36 Overall Well-being Subscale
Description: Use the SF-36 scale to measure the overall well-being from baseline to 6th month follow-up. Higher score indicates more peaceful, happy, and calm. Range (0-100)
Time Frame: Baseline and 6th month
Population: Some participants did not complete the questionnaire. 149 participants from PRISM B and 149 from PRISM C contributed to at least one of the two time points.
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 149 | 149
units in scale
  Baseline | 78.17 (16.1) | 80.38 (18.2)
  6th month follow-up: number analyzed (Participants) | 110 | 132
  6th month follow-up | 77.60 (18.2) | 82.12 (16.8)

4. Primary Outcome: Change in Social Isolation Measured by Friendship Scale
Description: Measures the level of social isolation from baseline to 12th month follow-up. Lower score means less social isolation. Range (0-24) .
Time Frame: Baseline and 12th month
Population: Some participants did not complete the questionnaire. 149 participants from PRISM B and 150 from PRISM C contributed to at least one of the two time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 149 | 150
units on a scale
  Baseline | 18.75 (4.1) | 19.72 (3.7)
  12th month follow-up: number analyzed (Participants) | 114 | 130
  12th month follow-up | 19.50 (3.9) | 20.24 (3.6)

5. Primary Outcome: Change in Level of Social Support Measured by Social Support Scale
Description: Measures the level of social support from baseline to 12th month follow-up. Higher score means more social support. Range (6-36).
Time Frame: Baseline and 12th month
Population: Some participants did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 150 | 150
units on a scale
  Baseline | 24.90 (6.9) | 25.33 (6.9)
  12th month follow-up: number analyzed (Participants) | 115 | 130
  12th month follow-up | 25.66 (7.00) | 26.55 (7.2)

6. Primary Outcome: Change Overall Well-being Measured by SF-36 Overall Well-being Subscale
Description: Use the SF-36 to measure the overall well-being from baseline to 12th month follow-up. Higher score means more peaceful, happy and calm. Range (0-100).
Time Frame: Baseline and 12th month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 149 | 149
units in scale
  Baseline | 78.17 (16.1) | 80.38 (18.2)
  12th month follow-up: number analyzed (Participants) | 111 | 130
  12th month follow-up | 75.78 (17.8) | 76.43 (19.6)

7. Secondary Outcome: Change in Computer Comfort Measured by Computer Attitude - Comfort Subscale .
Description: Use the computer attitude scale to measure the level of computer comfort from baseline to 6th month follow-up. Higher score means more computer comfort. Range (5-25).
Time Frame: baseline and 6 months
Population: Some participants did not complete the questionnaire. 148 participants from PRISM B and 149 from PRISM C contributed to at least one of the two time points.
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 149
units in scale
  Baseline | 16.64 (4.2) | 16.74 (4.2)
  6th month follow-up: number analyzed (Participants) | 109 | 132
  6th month follow-up | 16.45 (4.1) | 18.32 (4.5)

8. Secondary Outcome: Changes in Technology Proficiency Measured by Technology Proficiency Scale
Description: Measures the level of technology proficiency from baseline to 6th month follow-up. Higher scores means more computer proficiency. Range (6-30)
Time Frame: baseline and 6 months
Population: Some participants did not complete the questionnaire. 148 participants from PRISM B and 147 from PRISM C contributed to at least one of the two time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 147
units on a scale
  Baseline | 10.31 (4.7) | 9.87 (4.1)
  6th month follow-up: number analyzed (Participants) | 110 | 128
  6th month follow-up | 11.56 (5.0) | 17.65 (4.0)

9. Secondary Outcome: Change in Technology Adoption Measured by Technology Acceptance Questionnaire
Description: Measure the level of technology adoption from baseline to 6th month follow-up. Higher score means more acceptance. Range (6-42)
Time Frame: baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 149 | 149
units on a scale
  Baseline | 34.76 (7.4) | 34.70 (7.4)
  6th month follow-up: number analyzed (Participants) | 111 | 132
  6th month follow-up | 33.14 (8.2) | 32.82 (7.1)

10. Secondary Outcome: Change in Computer Comfort Measured by Computer Attitude - Comfort Subscale .
Description: Use the computer attitude scale to measure the level of computer comfort from baseline to 12th month follow-up. Higher score means more computer comfort. Range (5-25)
Time Frame: baseline and 12 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 149
units in scale
  Baseline | 16.64 (4.2) | 16.74 (4.2)
  12th month follow-up: number analyzed (Participants) | 113 | 128
  12th month follow-up | 16.35 (3.8) | 18.87 (4.5)

11. Secondary Outcome: Changes in Technology Proficiency Measured by Technology Proficiency Scale
Description: Measures the level of technology proficiency from baseline to 12th month follow-up. A higher score means more computer proficiency. Range (6-30)
Time Frame: baseline and 12 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 147
units on a scale
  Baseline | 10.31 (4.7) | 9.87 (4.1)
  12th month follow-up: number analyzed (Participants) | 113 | 126
  12th month follow-up | 11.44 (5.1) | 18.42 (4.6)

12. Secondary Outcome: Change in Technology Adoption Measured by Technology Acceptance Questionnaire
Description: Measures the level of technology adoption from baseline to 12th month follow-up. Higher score means more acceptance. Range (6-42)
Time Frame: baseline and 12 months
Population: Some participants did not answer the questionnaire. 149 participants from PRISM B and 149 from PRISM C contributed to at least one of the two time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 149 | 149
units on a scale
  Baseline | 34.76 (7.4) | 34.70 (7.4)
  12th month follow-up: number analyzed (Participants) | 112 | 128
  12th month follow-up | 33.22 (7.6) | 32.28 (8.0)

13. Secondary Outcome: Change in Computer Interest Measured by Computer Attitude - Interest Subscale
Description: Use the computer attitude scale to measure the level of computer interest from baseline to 6th month follow-up. Higher score means more interest towards computer. Range (5-25)
Time Frame: Baseline and 6th month follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 149
units in scale
  Baseline | 20.60 (3.2) | 20.46 (3.4)
  6th month follow-up: number analyzed (Participants) | 109 | 132
  6th month follow-up | 19.64 (3.8) | 21.20 (2.9)

14. Secondary Outcome: Change in Computer Interest Measured by Computer Attitude - Interest Subscale
Description: Use the computer attitude scale to measure the level of computer interest from baseline to 12th month follow-up. Higher score means more interest towards computer. Range (5-25)
Time Frame: Baseline and 12th month follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 149
units in scale
  Baseline | 20.60 (3.2) | 20.46 (3.4)
  12th month follow-up: number analyzed (Participants) | 113 | 127
  12th month follow-up | 19.94 (3.4) | 21.07 (3.2)

15. Secondary Outcome: Change in Computer Efficacy Measured by Computer Attitude - Efficacy Subscale
Description: Use the computer attitude scale to measure the level of computer efficacy from baseline to 12th month follow-up. Higher score means more efficacy towards computer. Range (5-25)
Time Frame: Baseline and 6th month follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 149
units in scale
  Baseline | 20.21 (3.2) | 20.30 (2.9)
  6th month follow-up: number analyzed (Participants) | 109 | 132
  6th month follow-up | 19.62 (3.4) | 21.02 (2.7)

16. Secondary Outcome: Change in Computer Efficacy Measured by Computer Attitude - Efficacy Subscale
Description: as for outcome 15
Time Frame: Baseline and 12th month follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units in scale
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Number analyzed (Participants) | 148 | 149
units in scale
  Baseline | 20.21 (3.2) | 20.3 (2.90)
  12th month follow-up: number analyzed (Participants) | 113 | 127
  12th month follow-up | 19.68 (3.3) | 20.83 (3.0)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not including serious) Adverse Events were not monitored/assessed.
Arm/Group | PRISM B: Notebook Condition | PRISM C: Computer Condition
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No